CLINICAL TRIAL: NCT07141537
Title: Caloric Balance Markers (CaBooM) Study
Brief Title: Caloric Balance Markers Study
Acronym: CaBooM
Status: Recruiting | Type: Observational
Sponsor: Institute for Systems Biology (Other)
Responsible Party: Sponsor
Other Study IDs: 2025.0037
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CaBooM: healthy adults

SUMMARY:
The purpose of CaBooM is to identify and characterize biomarkers of caloric balance-the relationship between energy intake (calories consumed) and energy expenditure (calories burned).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Able to travel to ISB for study visits.
* Able to read and communicate in English.

Exclusion Criteria:

* - Unable to provide informed consent.
* Is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2033-08-31 (Estimated); Study Completion 2033-08-31 (Estimated)

PRIMARY OUTCOMES:
caloric balance | 48 hours
  calories

CONTACTS AND LOCATIONS:
Overall Officials: Jared C Roach, MD, PhD, Principal Investigator — Institute for Systems Biology
Locations (1):
- Institute for Systems Biology, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No